CLINICAL TRIAL: NCT04555655
Title: Trial of A Chicken Extract and Peptide Supplement for the Prevention of Cognitive Decline and Mechanisms of Action in Non-demented Elderly Adults: A Multicenter, Two-year, Three-arm, Randomized, Double-blind, Placebo-controlled Study
Brief Title: The Effects of Chicken Extract and a Peptide Supplement for the Prevention of Cognitive Decline in Non-demented Elderly Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brand's Suntory Asia (Industry)
Collaborators: Taipei Medical University Shuang Ho Hospital (Other); National Cheng-Kung University Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BEC-CMI-003
Record Dates: First submitted 2020-09-03; First posted 2020-09-21 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-01

CONDITIONS: Cognitive Decline; Mild Cognitive Impairment; Aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chicken extract supplement (Experimental)
  Interventions: Dietary Supplement: Chicken extract supplement
- Peptides supplement (Experimental)
  Interventions: Dietary Supplement: Peptide Supplement
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Chicken extract supplement — 70ml of chicken extract supplement to be consumed daily in the morning before meals for 2 years.
  Arms: Chicken extract supplement
Dietary Supplement: Peptide Supplement — 70ml of Peptide Supplement (670mg) to be consumed daily in the morning before meals for 2 years.
  Arms: Peptides supplement
Other: Placebo — 70ml of placebo (caesinate) to be consumed daily in the morning before meals for 2 years.
  Arms: Placebo

SUMMARY:
This trial investigates the effect of a chicken extract supplement and a peptide supplement on cognitive function and potential mechanisms of action of cognitive decline during ageing, among non-demented elderly adults using a three-arm, randomized, placebo-controlled clinical trial design.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at 55 - 75 years of age
* Baseline cognition:
* Normal cognition with feelings of cognitive decline (subjective cognitive decline) OR
* Mild cognitive impairment (MCI+) with memory impairment
* Agree to participate in the study and provide written informed consent

Exclusion Criteria:

* Inadequate visual and auditory acuity to allow neuropsychological testing
* Significant cerebrovascular disease
* History of allergy to chicken meat
* Diagnosis of Alzheimer's disease (AD) with dementia or any other dementia
* Clinical dementia rating (CDR) score of > 0.5 at screening
* Evidence of other neurological, psychiatric or physical illness that can produce cognitive deterioration per investigator's judgment
* Inability or unwillingness to undergo PET scan
* Current diagnosis or history of alcoholism or substance addiction
* Regular use of any medication in the past 6 months that may affect cognitive functioning
* Regular use of cognitive enhancing supplements in the past 6 months
* Subjects with excessive blood donation or blood drawn prior to baseline
* Persons with a history of cardiovascular disease or any other cardiovascular or cerebrovascular diseases which investigators deem unsuitable to participate in the clinical study.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Cognitive Function assessed by Alzheimer's Disease Composite Score (ADCOMS) | 24 months
  Change from baseline in Alzheimer's Disease Composite Score (ADCOMS).
  ADCOMS composite score is a weighted linear combination of the 12 items in the Wold's partial least squares (PLS) model. Composite scores range from 0.0 to a maximum of 1.97, where higher values indicate worse performance.
Florbetaben (18F) PET Scan Imaging | 24 months
  Change from baseline values in Florbetaben (18F) PET scan

SECONDARY OUTCOMES:
Handgrip strength | 12 months & 24 months
  Change from baseline in handgrip strength
Ratio of plasma tau protein and amyloid-beta 42 | 24 months
  Change from baseline in plasma tau protein & amyloid-beta 42 ratio
Alzheimer's Disease Composite Score (ADCOMS) | 12 months
  Change from baseline in Alzheimer's Disease Composite Score (ADCOMS). ADCOMS composite score is a weighted linear combination of the 12 items in the Wold's partial least squares (PLS) model. Composite scores range from 0.0 to a maximum of 1.97, where higher values indicate worse performance.
Blood myeloperoxidase (MPO) levels | 12 months & 24 months
  Change from baseline in blood myeloperoxidase (MPO) Higher levels of MPO indicate worse oxidative stress status
Blood inflammation biomarker levels (hs-CRP, ESR, TNF-α, IL-6) | 12 months & 24 months
  Change from baseline in inflammation, measured by the following blood biomarkers. Each biomarker will be evaluated individually.
  1. High-sensitivity C-reactive Protein (hs-CRP)
  2. Erythrocyte Sedimentation Rate (ESR)
  3. Tumor necrosis factor alpha (TNFα)
  4. Interleukin 6 (IL-6)
Fasting blood glucose level | 4, 8, 12, 18 and 24 months
  Change from baseline in fasting blood glucose level
Taiwanese Depression Questionnaire (TQD) score | 4, 8, 12, 18 and 24 months
  Change from baseline in patient-reported Taiwanese Depression Questionnaire (TQD) scores.
  TDQ scores range from 0 to 54, with the higher score indicating the greater depression state.
Short Form-36 (SF-36) Component and Scale Scores | 4, 8, 12, 18 and 24 months
  Change from baseline in Short Form-36 (SF-36) Component and Scale Scores. Each scale is directly transformed into a 0 - 100 scale on the assumption that each question carries equal weight. Lower score indicates more disability/worse health status.
Athens Insomnia Scale (AIS) | 4, 8, 12, 18 and 24 months
  Change from baseline in Athens Insomnia Scale Score. A composite score which ranges from 0-24 will be evaluated. Higher score stands for greater severity of insomnia.
Incidence of infections | 24 months, reported at each study visit (4, 8, 12, 18 and 24 months)
  Number and incidence of infections occurring during the study period according to a self-reported infection survey
Cerebral blood flow measured with sonography | 12 months & 24 months
  Mean values of cerebral blood flow measured with sonography
Blood pressure (systolic blood pressure and diastolic blood pressure) | 4, 8, 12, 18 and 24 months
  Change from baseline in systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Taipei Medical University Hospital Shuang Ho Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - Taoyuan Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No